CLINICAL TRIAL: NCT06808503
Title: Implementing the NIMH Clinical Pathway in Rural Appalachian School-based Health Clinics
Brief Title: NIMH Clinical Pathway in Rural Appalachian School-based Health Clinics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Mary Christensen, Associate Professor and MSW Program Director, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2405972188
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Suicide Prevention; Suicide
MeSH Terms: conditions — Suicide Prevention; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): Review all medical records for patients for the standard of care used at the facility for suicide assessment and risk. Determine if the enrolled patients were assessed and if risks are present.
- NIMH Clinical Pathway (Active Comparator): Implementation of an adapted/tailored version of the NIMH Clinical Pathway, which identifies a workflow and tools for routine suicide risk screening, assessment, safety planning and follow-up.
  Interventions: Behavioral: NIMH Clinical Pathway

INTERVENTIONS:
Behavioral: NIMH Clinical Pathway — Complete the implemented workflow and tools for suicide risk screening, assessment, safety planning and follow-up.
  Arms: NIMH Clinical Pathway

SUMMARY:
This study will adapt and evaluate an evidence-based suicide risk screening and follow-up program in two school-based health centers in West Virginia. The suicide screening program is titled the "NIMH Clinical Pathway" and provides tools and procedures for routinely screening adolescents for suicide risk, completing risk assessments, safety planning, lethal means restriction, follow-up referrals, and other disposition planning as appropriate.

Investigators aim to do the following:

1. Gather formative data from providers, parents, and youth to inform ways to adapt and implement the NIMH Clinical Pathway so that it can be effectively implemented in rural, Appalachian School-Based Health Centers (SBHCs).
2. Gather preliminary data regarding the feasibility, acceptability, and effectiveness of the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Youth who are receiving services at the school-based health centers to participate
* Parents must be able to give legal consent for themselves and their children to participate
* Youth and Parent must be English-speaking
* Youth must also be able to give signed assent to participate
* Youth must be cognitively and medically able to participate in study activities

Exclusion Criteria:

* Youth in state custody will be excluded from study participation due to challenges related to obtaining legal consent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Screened for Suicidal Risks-Site 1 | Total period of 3 Months
  Review of patient records for the number of patients that were asked about suicidal thoughts and/or behaviors during their visit. Review will occur for a total of 3 months during the Treatment as Usual Period.
Number of Patients Screened for Suicidal Risks-Site 2 | Total period of 6 Months
  Review of patient records for the number of patients that were asked about suicidal thoughts and/or behaviors during their visit. Review will occur for a total of 6 months during the Treatment as Usual Period.
Number of Patients Reporting Suicidal Risks-Site 1 | Total period of 6 Months
  Review of patient records for the number of patients that reported having suicidal thoughts and/or behaviors. Review will occur for a total of 3 months during the Intervention Period.
Number of Patients Reporting Suicidal Risks-Site 2 | Total period of 3 Months
  Review of patient records for the number of patients that reported having suicidal thoughts and/or behaviors. Review will occur for a total of 6 months during the Interventional Period

SECONDARY OUTCOMES:
Safety Planning Rates (Number)- Site 1 | Initial Visit
  Number of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Number)- Site 1 | 3 Month Follow Up Visit
  Number of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Number)- Site 2 | Initial Visit
  Number of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Number)- Site 2 | 3 Month Follow Up Visit
  Number of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Percentage)- Site 1 | Initial Visit
  Percentage of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Percentage)- Site 2 | Initial Visit
  Percentage of at-risk patients that the providers documented safety planning was completed.
Safety Planning Rates (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of at-risk patients that the providers documented safety planning was completed.
Follow-up Service Provision (Number)- Site 1 | Chart review conducted within 3 months following initial visit
  Number of at-risk patients that documentation confirms providers conducted follow-up appointments to re-assess suicidal symptoms.
Follow-up Service Provision (Number)- Site 2 | Chart review conducted within 3 months following initial visit
  Number of at-risk patients that documentation confirms providers conducted follow-up appointments to re-assess suicidal symptoms.
Participant rate of Suicidal Ideation: (SIQ-Jr)- Site 1 | Initial Visit
  Suicidal Ideation Questionnaire (SIQ-Jr) will be administered to participants at the initial visit and 3 months follow up. The SIQ-Jr is a 15-item self-report questionnaire that measures suicidal thoughts on a 7-point scale ("0- I never had this thought" to "6- I have this thought every day"). Scores range from 0-90, SIQ-Jr scores of 23 and above indicate severe suicidal ideation and the need for clinical intervention.
Participant rate of Suicidal Ideation: (SIQ-Jr)- Site 1 | 3 Month Follow Up Visit
  Suicidal Ideation Questionnaire (SIQ-Jr) will be administered to participants at the initial visit and 3 months follow up. The SIQ-Jr is a 15-item self-report questionnaire that measures suicidal thoughts on a 7-point scale ("0- I never had this thought" to "6- I have this thought every day"). Scores range from 0-90, SIQ-Jr scores of 23 and above indicate severe suicidal ideation and the need for clinical intervention.
Participant rate of Suicidal Ideation: (SIQ-Jr)- Site 2 | Initial visit
  Suicidal Ideation Questionnaire (SIQ-Jr) will be administered to participants at the initial visit and 3 months follow up. The SIQ-Jr is a 15-item self-report questionnaire that measures suicidal thoughts on a 7-point scale ("0- I never had this thought" to "6- I have this thought every day"). Scores range from 0-90, SIQ-Jr scores of 23 and above indicate severe suicidal ideation and the need for clinical intervention.
Participant rate of Suicidal Ideation: (SIQ-Jr)- Site 2 | 3 Month Follow Up Visit
  Suicidal Ideation Questionnaire (SIQ-Jr) will be administered to participants at the initial visit and 3 months follow up. The SIQ-Jr is a 15-item self-report questionnaire that measures suicidal thoughts on a 7-point scale ("0- I never had this thought" to "6- I have this thought every day"). Scores range from 0-90, SIQ-Jr scores of 23 and above indicate severe suicidal ideation and the need for clinical intervention.
Participant rate of Depression: (CES-D)- Site 1 | Initial Visit
  The Center for Epidemiological Studies Depression Scale (CES-D) will be administered to the participant at the initial visit and the 3 month follow up. The CES-D is a self-report measure with 10 items asking about the frequency with which individuals have experienced various symptoms of depression within the last week. Each item is rated on a Likert scale, typically ranging from 0 (rarely or none of the time) to 3 (most or all of the time). Total scores range is from 0-30, with higher scores indicating higher levels of depression.
Participant rate of Depression: (CES-D)- Site 1 | 3 Month Follow Up Visit
  The Center for Epidemiological Studies Depression Scale (CES-D) will be administered to the participant at the initial visit and the 3 month follow up. The CES-D is a self-report measure with 10 items asking about the frequency with which individuals have experienced various symptoms of depression within the last week. Each item is rated on a Likert scale, typically ranging from 0 (rarely or none of the time) to 3 (most or all of the time). Total scores range is from 0-30, with higher scores indicating higher levels of depression.
Participant rate of Depression: (CES-D)- Site 2 | Initial Visit
  The Center for Epidemiological Studies Depression Scale (CES-D) will be administered to the participant at the initial visit and the 3 month follow up. The CES-D is a self-report measure with 10 items asking about the frequency with which individuals have experienced various symptoms of depression within the last week. Each item is rated on a Likert scale, typically ranging from 0 (rarely or none of the time) to 3 (most or all of the time). Total scores range is from 0-30, with higher scores indicating higher levels of depression.
Participant rate of Depression: (CES-D)- Site 2 | 3 Month Follow Up Visit
  The Center for Epidemiological Studies Depression Scale (CES-D) will be administered to the participant at the initial visit and the 3 month follow up. The CES-D is a self-report measure with 10 items asking about the frequency with which individuals have experienced various symptoms of depression within the last week. Each item is rated on a Likert scale, typically ranging from 0 (rarely or none of the time) to 3 (most or all of the time). Total scores range is from 0-30, with higher scores indicating higher levels of depression.
Participants with Suicidal Behavior at Follow Up (Number)- Site 1 | 3 Month Follow Up Visit
  Number of participants who indicate "yes" as per the following: Providers will administer the brief version of the Columbia Suicide-Severity Rating Scale (C-SSRS). The C-SSRS is a screening tool that asks two initial questions about suicidal ideation. For participants who state "yes" to either of these questions, they are asked additional questions about suicidal intent, plans, and behavior. Investigators will measure suicidal behavior as a dichotomous "yes"/"no" variable. A participant will be considered a "yes" for this measure if they answer "yes" to the final question about engaging in suicidal preparation and/or attempts on the C-SSRS and to the question asking whether or not they have done so in the past 3 months.
Participants with Suicidal Behavior at Follow Up (Number)- Site 2 | 3 Month Follow Up Visit
  Number of participants who indicate "yes" as per the following: Providers will administer the brief version of the Columbia Suicide-Severity Rating Scale (C-SSRS). The C-SSRS is a screening tool that asks two initial questions about suicidal ideation. For participants who state "yes" to either of these questions, they are asked additional questions about suicidal intent, plans, and behavior. Investigators will measure suicidal behavior as a dichotomous "yes"/"no" variable. A participant will be considered a "yes" for this measure if they answer "yes" to the final question about engaging in suicidal preparation and/or attempts on the C-SSRS and to the question asking whether or not they have done so in the past 3 months.
Participants with Suicidal Behavior at Follow Up (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of participants who indicate "yes" as per the following: Providers will administer the brief version of the Columbia Suicide-Severity Rating Scale (C-SSRS). The C-SSRS is a screening tool that asks two initial questions about suicidal ideation. For participants who state "yes" to either of these questions, they are asked additional questions about suicidal intent, plans, and behavior. Investigators will measure suicidal behavior as a dichotomous "yes"/"no" variable. A participant will be considered a "yes" for this measure if they answer "yes" to the final question about engaging in suicidal preparation and/or attempts on the C-SSRS and to the question asking whether or not they have done so in the past 3 months.
Participants with Suicidal Behavior at Follow Up (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of participants who indicate "yes" as per the following: Providers will administer the brief version of the Columbia Suicide-Severity Rating Scale (C-SSRS). The C-SSRS is a screening tool that asks two initial questions about suicidal ideation. For participants who state "yes" to either of these questions, they are asked additional questions about suicidal intent, plans, and behavior. Investigators will measure suicidal behavior as a dichotomous "yes"/"no" variable. A participant will be considered a "yes" for this measure if they answer "yes" to the final question about engaging in suicidal preparation and/or attempts on the C-SSRS and to the question asking whether or not they have done so in the past 3 months.
Participants Reporting Safety Plan Usage (Number) - Site 1 | 3 Month Follow Up Visit
  Number of participants who screen positive for suicide risk during the initial visit reporting use of the safety plan developed for the participant.
Participants Reporting Safety Plan Usage (Number)- Site 2 | 3 Month Follow Up Visit
  Number of participants who screen positive for suicide risk during the initial visit reporting use of the safety plan developed for the participant.
Participants Reporting Safety Plan Usage (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of participants who screen positive for suicide risk during the initial visit reporting use of the safety plan developed for the participant.
Participants Reporting Safety Plan Usage (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of participants who screen positive for suicide risk during the initial visit reporting use of the safety plan developed for the participant.
Parents Reporting Safety Plan Usage (Number)- Site 1 | 3 Month Follow Up Visit
  Number of parents whose child screened positive for suicide risk during the initial visit reporting the use of the safety plan that was developed for the participant (child).
Parents Reporting Safety Plan Usage (Number)- Site 2 | 3 Month Follow Up Visit
  Number of parents whose child screened positive for suicide risk during the initial visit reporting the use of the safety plan that was developed for the participant (child).
Parents Reporting Safety Plan Usage (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of parents whose child screened positive for suicide risk during the initial visit reporting the use of the safety plan that was developed for the participant (child).
Parents Reporting Safety Plan Usage (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of parents whose child screened positive for suicide risk during the initial visit reporting the use of the safety plan that was developed for the participant (child).
Participants Reporting Frequency of Safety Plan Use (Number)- Site 1 | 3 Month Follow Up Visit
  Number of participants who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Participants Reporting Frequency of Safety Plan Use (Number)- Site 2 | 3 Month Follow Up Visit
  Number of participants who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Participants Reporting Frequency of Safety Plan Use (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of participants who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Participants Reporting Frequency of Safety Plan Use (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of participants who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Parents Reporting Frequency of Safety Plan Use (Number)- Site 1 | 3 Month Follow Up Visit
  Number of parents who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Parents Reporting Frequency of Safety Plan Use (Number)- Site 2 | 3 Month Follow Up Visit
  Number of parents who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Parents Reporting Frequency of Safety Plan Use (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of parents who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Parents Reporting Frequency of Safety Plan Use (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of parents who endorse each category related to Safety Plan Usage. Measured on a Likert Type scale with a range of 1-5 ("1-all the time," "2-often," "3-sometimes," "4-almost never," or "5-never") with 1 being more frequent usage and 5 being less frequent usage.
Participants Reporting Helpfulness of Safety Plan (Number)- Site 1 | 3 Month Follow Up Visit
  Number of participants who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Participants Reporting Helpfulness of Safety Plan (Number)- Site 2 | 3 Month Follow Up Visit
  Number of participants who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Participants Reporting Helpfulness of Safety Plan (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of participants who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Participants Reporting Helpfulness of Safety Plan (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of participants who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Parents Reporting Helpfulness of Safety Plan (Number)- Site 1 | 3 Month Follow Up Visit
  Number of parents who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Parents Reporting Helpfulness of Safety Plan (Number)- Site 2 | 3 Month Follow Up Visit
  Number of parents who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Parents Reporting Helpfulness of Safety Plan (Percentage)- Site 1 | 3 Month Follow Up Visit
  Percentage of parents who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Parents Reporting Helpfulness of Safety Plan (Percentage)- Site 2 | 3 Month Follow Up Visit
  Percentage of parents who endorse each category related to Safety Plan Helpfulness. Measured on a Likert Type scale with a range of 1-4 ("1-very helpful," "2-helpful," "3-a little helpful," or "4-not at all helpful.") with 1 being most helpful and 4 being least helpful.
Participants Reporting Acute Care Usage (Number)- Site 1 | Total period of 3 Months
  Number of participants who report acute care was utilized for help with suicidal symptoms between the initial visit and the 3 month follow up visit per participant report.
Participants Reporting Acute Care Usage (Number)- Site 2 | Total period of 3 Months
  Number of participants who reported acute care was utilized for help with suicidal symptoms between the initial visit and the 3 month follow up visit per participant report.
Participants Reporting Acute Care Usage (Percentage)- Site 1 | Total period of 3 Months
  Percentage of participants that reported acute care was utilized for help with suicidal symptoms between the initial visit and the 3 month follow up visit.
Participants Reporting Acute Care Usage (Percentage)- Site 2 | Total period of 3 Months
  Percentage of participants that reported acute care was utilized for help with suicidal symptoms between the initial visit and the 3 month follow up visit.
Parents Reporting Acute Care Usage (Number)- Site 1 | Total period of 3 Months
  Number of parents who report a participant utilized acute care for help with suicidal symptoms between the initial visit and the 3 month follow up visit as per reported by the parent.
Parents Reporting Acute Care Usage (Number)- Site 2 | Total period of 3 Months
  Number of parents who report a participant utilized acute care for help with suicidal symptoms between the initial visit and the 3 month follow up visit as per reported by the parent.
Parents Reporting Acute Care Usage (Percentage)- Site 1 | Total period of 3 Months
  Percentage of parents that reported acute care was utilized for help with participant suicidal symptoms between the initial visit and the 3 month follow up visit.
Parents Reporting Acute Care Usage (Percentage)- Site 2 | Total period of 3 Months
  Percentage of parents that reported acute care was utilized for help with participant suicidal symptoms between the initial visit and the 3 month follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Christensen, PhD, LICSW, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No